CLINICAL TRIAL: NCT03512067
Title: Entrainment-Based Mechanical Ventilation to Improve Patient-Ventilator Synchrony
Brief Title: Entrainment-Based Mechanical Ventilation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative reasons and Overall Study PI moved to another institution.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Gyorgy Frendl, M.D., Ph.D., Associate Professor, Director of Surgical Critical Care Research, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013P001506; 5R34HL125859-02 (NIH)
Record Dates: First submitted 2018-04-11; First posted 2018-04-30 (Actual); Results first posted 2019-08-28 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Respiratory Insufficiency; Respiratory Failure; Mechanical Ventilation Complication
Keywords: Mechanical Ventilation; Respiratory Support
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: This study is a device trial to examine the efficacy of the new mode of mechanical ventilation. It will be single-armed and open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Patients given EMV Ventilation (Experimental): Baseline mechanical ventilation data with conventional pressure-limited assist/control ventilation mode will then be collected for a 4-hour period. The patients will then be transitioned to pressure-limited entrainment-based ventilation for a 4-hour period. Baseline ventilation monitoring will be carried out either immediately preceding or immediately following EMV in the same patient. The sequence of the control/baseline phase and the experimental phase of the study will be randomized.
  Interventions: Device: Patients given EMV Ventilation

INTERVENTIONS:
Device: Patients given EMV Ventilation — Baseline mechanical ventilation data with conventional pressure-limited assist/control ventilation mode will then be collected for a 4-hour period. The patients will then be transitioned to pressure-limited entrainment-based ventilation for a 4-hour period. Baseline ventilation monitoring will be carried out either immediately preceding or immediately following EMV in the same patient. The sequence of the control/baseline phase and the experimental phase of the study will be randomized.

SUMMARY:
BACKGROUND AND SIGNIFICANCE Entrainment-based ventilation is a new mode of mechanical ventilation based on the classical physics theory of mutual entrainment between coupled oscillators. Typically, the entrained inspiratory activity may precede or lag behind machine inflation depending on whether spontaneous respiratory frequency is higher or lower than the ventilator frequency.

HYPOTHESIS The investigators anticipate that the results of the study will help to improve the interaction of patients with the mechanical ventilator thereby minimizing the risks of mechanical ventilation in future. The investigators believe the potential benefits significantly outweigh the potential risks.

RESEARCH STUDY DESIGN AND METHODS This is a prospective study and single site. Twenty mechanically ventilated patients, stable on their current vent settings and are capable of triggering the ventilator in the SICU, MICU, CCU and Cardiac and Neuro Surgery ICUs at BWH will be recruited.

After obtaining informed consent a respiratory real-time data monitor will be placed between the artificial airway and the Y piece of the ventilator circuit. Baseline mechanical ventilation data with conventional pressure-limited assist/control ventilation mode will then be collected for a 4-hour period. The patients will then be transitioned to pressure-limited entrainment-based ventilation for a 4-hour period. Baseline ventilation monitoring will be carried out either immediately preceding or immediately following EMV in the same patient. The sequence of the control/baseline phase and the experimental phase of the study will be randomized.

DATA COLLECTION Demographic data, weight, height, and past and current medical history will be recorded. Also hospital admission information, reasons of mechanical ventilation, mode of mechanical ventilation and settings, arterial blood gas, clinical laboratory (hematology/chemistry) values, and hemodynamic values will be recorded.

STATISTICAL ANALYSIS Baseline demographic and procedural variables will be analyzed statistically by plotting the 95% confidence intervals of each variable. For feasibility evaluation, the total number of each type of asynchronous breaths/hour during entrainment-based ventilation will be averaged over the 4-hour experimental period and compared with those in the 4-hour baseline ventilation period.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE

All currently available mechanical ventilation modes assume that patient-ventilator interaction is necessarily a "master-slave" or controller-follower relationship. In controlled mechanical ventilation, the ventilator takes control of the ventilatory rhythm irrespective of whether the patient is breathing or not. In the patient-triggered mechanical ventilation modes such as assist/control, pressure support ventilation, proportional assist ventilation, neutrally adjusted ventilator support), instead of the ventilator dictating the ventilatory rhythm (ventilator-based ventilation), patient triggering allows the patient to initiate the breath with the ventilator responding to the patients demand (patient-based ventilation) with the imposition of various support.

Entrainment-based mechanical ventilation (EMV) is a new mode of mechanical ventilation based on the classical physics theory of mutual entrainment between coupled oscillators. It takes advantage of the patient's powerful innate capacity to entrain 1:1 to the ventilator rhythm via the Herring-Breuer reflex, provided that the ventilator rhythm is close enough to the spontaneous breathing rhythm. This ability of the respiratory system to adapt to changes in the entrainment mechanism via habituation and desensitization of the Herring-Breuer reflex allows an even greater dynamic range of entrainment.

Justification for the investigation

The investigators anticipate that the results of the study will help to improve the interaction of patients with the mechanical ventilator thereby minimizing the risks of mechanical ventilation in future. We believe the potential benefits significantly outweigh the potential risks.

METHODS

This is a prospective study designed to evaluate the ability of entrainment-based mechanical ventilation to provide synchronous mechanical ventilation to patients in the SICU, MICU, CCU and Cardiac and Neuro Surgery ICUs at the Brigham and Women's Hospital (BWH).

Study design and procedures:

After obtaining informed consent a respiratory real-time data monitor will be placed between the artificial airway and the Y piece of the ventilator circuit. Baseline mechanical ventilation data with conventional pressure-limited assist/control ventilation mode will then be collected for a 4-hour period. The patients will then be transitioned to pressure-limited entrainment-based ventilation for a 4-hour period. Baseline ventilation monitoring will be carried out either immediately preceding or immediately following EMV in the same patient. The sequence of the control/baseline phase and the experimental phase of the study will be randomized.

During the observation study period, the basic ventilator settings will remain as prescribed during conventional mechanical ventilation. Any adjustment in basic ventilator settings will be up to the medical staff caring for the patient. Throughout the observational period a respiratory therapist familiar with the operation of entrainment-based ventilation will be at the patients' bedside constantly observing the patients interaction with the ventilator. In addition, the ventilator alarms and limits will be set appropriately preventing the airway pressure from increasing more than 5 cmH2O above the set level or the respiratory rate or tidal volume from exceeding or decreasing below the patient average tidal volume or respiratory rate by more than 25%. Apnea backup ventilation will be set to activate after a 20 second apnea period.

Data collection:

Demographic data, weight, height, and past and current medical history will be recorded. Also hospital admission information, reasons of mechanical ventilation, mode of mechanical ventilation and settings, arterial blood gas, clinical laboratory (hematology/chemistry) values, and hemodynamic values will be recorded.

A respiratory real-time data monitor will continuously collect mechanical ventilation data, which will be downloaded to a laptop computer for later analysis.

Blood gas analysis will be performed at the 2nd hr and at end of the baseline ventilation period, 2nd hr and at the end of the entrainment-based ventilation period.

Oxygen saturation and blood pressure will be recorded every 15 minutes (every 5 minutes in the first hour) until completion.

ECG will be monitored continuously and recorded every 15 minutes (every 5 minutes in the first hour).

Heart rate, paradoxical breathing, accessory muscle use, nasal flaring, will be continuously monitored throughout the study.

Safety criteria:

The following criteria will be used to identify failure of entrainment-based ventilation:

RR > 35/min for > 5 min SpO2 < 88% for 5 minutes and not corrected by suctioning or if SpO2 < 80% at any time Pulse sustained < 50/min or > 120/min PH + 0.05 units from baseline pH PCO2 + 10 mmHg from baseline PCO2 Mean arterial pressure sustained + 20 mmHg from baseline pressure Ischemic changes on ECG New onset of paradoxical breathing, accessory muscle use, nasal flaring, etc. Agitation (RASS > +1), diaphoresis, persistent anxiety despite reassurance and requiring sedation.

Once any of these safety criteria are met, the patient will be placed back to the baseline ventilation mode and closely observed for return to the pre-intervention baseline. Any patient who does not return to a pre-intervention baseline within 5 minutes after return to baseline ventilator settings will be evaluated by the study doctor for possible adverse effects or serious adverse effects and the patient will not be given further EMV therapy. Such AEs or SAEs will be deemed unknown related UADE or USADE. The DSMB will review the data and any safety concerns along with the Investigator and Sponsor each time any adverse event or serious adverse event occurs regardless of whether such an event is device related or not. If three or more non-serious adverse events occur or if two serious adverse events occur or if any death occurs, the corresponding events will be deemed possibly device related and the study will be placed on hold and the DSMB will review all available data at the time of the hold. The FDA and IRBs would review and approve any and all modifications to the protocol in response to such a study hold. Unanticipated problems and adverse events that occur during the conduct of the study, after study completion, or after subject withdrawal or completion will be reported to the IRB within 5 working days/7 calendar days of the date the investigator first becomes aware of the problem.

The first indications of any adverse events: such as bronchospasm, atelectasis, hypoxemia, barotraumas, pulmonary edema, prolonged mechanical ventilation, increased ventilatory requirements, pneumonia, pneumothorax, acute lung injury, ARDS, organ failure, MI, or death are abnormal cardiorespiratory responses meeting the above safety criteria will be reported to the IRB and FDA according to the guidelines. Serious adverse events will be defined as any of the previous adverse events that lead to death, or are life-threatening, or lead to persistent or significant disability/incapacity, prolongation of hospitalization or surgical procedures. Investigators will monitor all subjects for any adverse events or serious adverse events for 48 hours after return to baseline mechanical ventilation and will specifically include each of the above-listed events or any other adverse events or serious adverse events in the case report forms.

Patient monitoring:

This study will be performed at the subject's bedside when the subject is stable. A standard ventilator modified to provide entrainment-based ventilation will be used for the study. All ventilator alarms will be active.

During the study period a respiratory therapist and study staff will constantly monitor the patient for adverse or serious adverse events. If any of the events listed in the safety criteria above occurs, the entrainment-based ventilation will be permanently discontinued and subject will be changed back to baseline or conventional ventilation. Also the study will be stopped if any SAEs occur.

The protocol calls for blood gas analysis at the 2nd hr and at the end of the EMV period. Therefore, changes in arterial pH and PCO2 values from baseline will be assessed at those time intervals for any violation of the safety criteria. Once any changes in these blood gas variables are found to violate the stated safety criteria, the patient will be immediately returned to the pre-intervention ventilator settings and closely observed for return to the pre-intervention baseline.

ECG will be monitored continuously and recorded every 15 minutes (every 5 minutes in the first hour). Mean arterial pressure will be recorded every 15 minutes (every 5 minutes in the first hour).

Once any ischemic changes on ECG or excessive changes in mean arterial pressure (+ 20 mm Hg from baseline) are detected, the patient will be immediately returned to the pre-intervention ventilator settings and closely observed for return to the pre-intervention baseline.

For all other safety criteria mentioned above (regarding pulse, paradoxical breathing, accessory muscle use, nasal flaring, etc.), the timeframes are similar to those for RR. Specifically, the patient will be monitored continuously and will be placed back to the baseline mode of ventilation if any of these safety criteria are violated for > 5 min.

Sedation management will be performed per BWH ICU sedation guidelines, with sedation targeted to Ricker Agitation Sedation Scale.

Statistical analysis

Our study is targeted to enroll at least 20 sequential mechanically ventilated patients. Baseline demographic and procedural variables will be analyzed statistically by plotting the 95% confidence intervals of each variable. With 20 patients we will have an 88% chance of seeing any complication (such as those defined by the safety criteria or any associated adverse event or serious adverse event) that occurs with a frequency of 10% or more. For feasibility evaluation, the total number of each type of asynchronous breaths/hour during entrainment-based ventilation will be averaged over the 4-hour experimental period and compared with those in the 4-hour baseline ventilation period. The 95% confidence intervals of the differences of each type of asynchrony between entrainment-based ventilation and baseline ventilation will be provided without formal inference of statistical significance.

Analysis of synchrony:

The following types of patient-ventilator asynchrony will be analyzed every hour over the 4-hour baseline period and 4-hour experimental period:

Trigger asynchrony - Number of breaths/hour initiated by the patients that fail to trigger the ventilator to inspiration (identified by pressure, flow and or CO2 ventilator graphics.

Breath initiation asynchrony - Number of breaths/hour in which the initial airway pressure drops below baseline pressure for > 100 milliseconds prior to pressurization of the airway or a concave rise in airway pressure after triggering or an initial pressure increase that exceeds the set pressure level.

Breath termination asynchrony - Number of breaths/hour in which airway pressure at the end of the pressure targeted breath increases above set level just prior to exhalation or a second breath is rapidly triggered (double triggering) during initial expiration or premature termination of breath with small tidal volume.

Rhythm asynchrony - Number of breaths/hour in which ventilation is continuously patient-triggered (assist mode) or continuously ventilator-initiated (control mode) for more than 10 minutes.

Risk minimization

The EMV method is an extension of the well-established assist/control (A/C) ventilation mode and has minimal risk.

ELIGIBILITY:
Inclusion Criteria:

* Adult (at least 18 years of age), mechanically ventilated via endotracheal tube, of either sex
* Capable of triggering the ventilator
* Subject receiving pressure support ventilation (or assist/control pressure-limited mechanical ventilation) with less than or equal to 15 cm H2O inspiratory pressure, or, if on volume-limited A/C, when switched to pressure-limited A/C with the inspiratory pressure set to match the tidal volume on volume-limited A/C, the resultant inspiratory pressure is less than or equal to 15 cm H2O.
* Stable on the above-mentioned ventilatory support for at least 8 hours.
* Arterial line in place for obtaining arterial blood gases

Exclusion Criteria:

* Requiring high inspiratory oxygen concentration (> 50%).
* Requiring high ventilatory driving pressure (> 15 cm H20 on pressure-support)
* High spinal cord injury
* Immunosuppressed, < 2 months after receiving chemotherapy or radiation therapy.
* Neuromuscular/ neurological disease of a progressive nature resulting in chronic ventilator dependence.
* High risk of mortality within 3 months (terminal stage of their disease).
* Unable to spontaneously trigger the ventilator for any reason.
* Not considered a candidate for weaning from ventilatory support
* Consented for another interventional study.
* Requiring deep sedation and analgesia [Richmond Agitation Sedation Scale -3 to -5 (RASS)]
* Hemodynamically unstable patients as defined by those requiring norepinephrine at a dose greater than 5 mcg/min or neosynephrine > 100 mcg/min or those with a mean arterial blood pressure < 55 or > 120 mmHg or those with a heart rate < 50 or > 140 bpm.
* Respiratory rate > 30 breaths/min
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-09-02 (Actual); Study Completion 2018-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Sang Poon, PhD, Study Director — Massachusetts Institute of Technology; Gyorgy Frendl, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] MacDonald SM, Song G, Poon CS. Nonassociative learning promotes respiratory entrainment to mechanical ventilation. PLoS One. 2007 Sep 12;2(9):e865. doi: 10.1371/journal.pone.0000865. PMID 17848996
- [Background] Petrillo GA, Glass L, Trippenbach T. Phase locking of the respiratory rhythm in cats to a mechanical ventilator. Can J Physiol Pharmacol. 1983 Jun;61(6):599-607. doi: 10.1139/y83-092. PMID 6576843
- [Background] Muzzin S, Baconnier P, Benchetrit G. Entrainment of respiratory rhythm by periodic lung inflation: effect of airflow rate and duration. Am J Physiol. 1992 Aug;263(2 Pt 2):R292-300. doi: 10.1152/ajpregu.1992.263.2.R292. PMID 1510169
- [Background] Baconnier PF, Benchetrit G, Pachot P, Demongeot J. Entrainment of the respiratory rhythm: a new approach. J Theor Biol. 1993 Sep 21;164(2):149-62. doi: 10.1006/jtbi.1993.1145. PMID 8246514
- [Background] Vibert JF, Caille D, Segundo JP. Respiratory oscillator entrainment by periodic vagal afferentes: an experimental test of a model. Biol Cybern. 1981;41(2):119-30. doi: 10.1007/BF00335366. No abstract available. PMID 7248341
- [Background] Petrillo GA, Glass L. A theory for phase locking of respiration in cats to a mechanical ventilator. Am J Physiol. 1984 Mar;246(3 Pt 2):R311-20. doi: 10.1152/ajpregu.1984.246.3.R311. PMID 6584038
- [Background] Muzzin S, Trippenbach T, Baconnier P, Benchetrit G. Entrainment of the respiratory rhythm by periodic lung inflation during vagal cooling. Respir Physiol. 1989 Feb;75(2):157-72. doi: 10.1016/0034-5687(89)90060-1. PMID 2711050
- [Background] Graves C, Glass L, Laporta D, Meloche R, Grassino A. Respiratory phase locking during mechanical ventilation in anesthetized human subjects. Am J Physiol. 1986 May;250(5 Pt 2):R902-9. doi: 10.1152/ajpregu.1986.250.5.R902. PMID 3706575
- [Background] Simon PM, Zurob AS, Wies WM, Leiter JC, Hubmayr RD. Entrainment of respiration in humans by periodic lung inflations. Effect of state and CO(2). Am J Respir Crit Care Med. 1999 Sep;160(3):950-60. doi: 10.1164/ajrccm.160.3.9712057. PMID 10471624
- [Background] Simon PM, Habel AM, Daubenspeck JA, Leiter JC. Vagal feedback in the entrainment of respiration to mechanical ventilation in sleeping humans. J Appl Physiol (1985). 2000 Aug;89(2):760-9. doi: 10.1152/jappl.2000.89.2.760. PMID 10926663

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Given EMV Ventilation: Baseline mechanical ventilation data with conventional pressure-limited assist/control ventilation mode will then be collected for a 4-hour period. The patients will then be transitioned to pressure-limited entrainment-based ventilation (EMV) for a 4-hour period. Baseline ventilation monitoring will be carried out either immediately preceding or immediately following EMV in the same patient. The sequence of the control/baseline phase and the experimental phase of the study will be randomized.
Period: Overall Study
Arm/Group | Patients Given EMV Ventilation
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Given EMV Ventilation
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 60 [NA to NA] — Only 1 patient was enrolled in the study, so a full range cannot be given.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1
Respiratory Rate [Number; unit: breaths/minute] | 12

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Evaluation
Description: Total number of asynchronous breaths/hour during entrainment-based ventilation compared to baseline ventilation.
Time Frame: 8 Hours
Measure: Number; unit: breaths
Arm/Group | Patients Given EMV Ventilation
Number analyzed (Participants) | 1
breaths
  4 Hour Session 1: Total # of Asynchronous Breaths | 1372
  4 Hour Session 2: Total # of Asynchronous Breaths | 1402

2. Secondary Outcome: Assess for Frequency of Complications Related to the Use of EMV
Description: With 20 patients we will have an 88% chance of seeing any complication (such as those defined by the safety criteria or any associated adverse event or serious adverse event) that occurs with a frequency of 10% or more.
Time Frame: 8 Hours
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Given EMV Ventilation
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 month during the patient's length of stay at the hospital.
Arm/Group | Patients Given EMV Ventilation
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Early termination led to small numbers of subjects (only one participant) analyzed.

Study was terminated early due to administrative reasons and Overall Study PI (Dr. Chi-Sang Poon) moving to another institution

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT03512067/Prot_SAP_001.pdf